CLINICAL TRIAL: NCT00717028
Title: Achados da avaliação videoendoscópica da deglutição em crianças Com Paralisia Cerebral.
Brief Title: Functional Endoscopic Evaluation of Swallowing
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Responsible Party: Renata Cavalcante Barbosa Haguette, UNIFOR
Other Study IDs: 198/2005
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2005-09

CONDITIONS: Cerebral Palsy; Dysphagia
Keywords: Cerebral palsy; Dysphagia; Deglutition; Endoscopy
MeSH Terms: conditions — Cerebral Palsy; Deglutition Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators objective is to describe functional endoscopic evaluation of swallowing findings in children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a predominantly motor disorder and dysphagia is a frequent complaint. Functional endoscopic evaluation of swallowing (FESS) involves anatomic and functional observation of the larynx and pharynx, evaluation of swallowing and maneuvers to improve it, also testing the laryngeal sensitivity. We evaluated nine patients with CP of both sexes, which age varied from 1 to 10 years old, attended at dysphagia multidisciplinary clinic, at NAMI (Integrated Medical Assistance Nucleons).

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of cerebral palsy.

Exclusion Criteria:

* medical diagnoses not associated with cerebral palsy that affect swallowing.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Haguette, Mestre, Principal Investigator — Fortaleza University
Locations (1):
- Dysphagia multidisciplinary clinic at Integrated Medical Assistance Nucleons, Fortaleza, Ceará, Brazil